CLINICAL TRIAL: NCT06519864
Title: Validity and Reliability of a Novel Depth Camera-based Physical Function and Fall Risk Assessments for Community Dwellings Elders Living Alone
Brief Title: Validity and Reliability of a Depth Camera-based Automated Physical Function and Fall Risk Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Changho Song, Professor, Principal Investigator, Sahmyook University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: SYU 2022-06-003-005
Record Dates: First submitted 2024-07-08; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Fall; Healthy Aging
MeSH Terms: interventions — Hand Strength

STUDY DESIGN:
Intervention Model Description: A cross-sectional design
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elders over 65-year-old (Experimental): * Those who are elders (≥65 years)
  * The enrolled participants completes the following evaluations during a single session: Tandem Stance Test (TST), Five Times Sit to Stand Test (FTSS), Turn Up and Go Test (TUG), Berg Balance Scale (BBS), Functional Reach Test (FRT), Four Square Step Test (FSST), Grip Strength (GS), and Short Physical Performance Battery (SPPB). The AK-based measurements are TST, FTSS, and TUG which are also the components of the SPPB.
  Interventions: Diagnostic Test: Azure Kinect-based Tandem Stance Test (ATST) and Physical Therapist's Measurements of Tandem Stance Test (PTST); Diagnostic Test: Azure Kinect-based Five Times Sit-to-Stand Test (AFTSS) and Physical Therapist's Measurements of Five Times Sit-to-Stand Test (PFTSS); Diagnostic Test: Azure Kinect-based Timed Up and Go Test (ATUG) and Physical Therapist's Measurements of Timed Up and Go Test (PTUG); Diagnostic Test: Short Physical Performance Battery (SPPB); Diagnostic Test: Berg Balance Scale (BBS); Diagnostic Test: Functional Reach Test (FRT); Diagnostic Test: Four-Square Step Test (FSST); Diagnostic Test: Grip Strength (GS)
- Healthy adults under 65-year-old (Active Comparator): * Those who are young adults over 18 and under 65 years old
  * The enrolled participants completes the following evaluations during a single session: Tandem Stance Test (TST), Five Times Sit to Stand Test (FTSS), Turn Up and Go Test (TUG), Berg Balance Scale (BBS), Functional Reach Test (FRT), Four Square Step Test (FSST), Grip Strength (GS), and Short Physical Performance Battery (SPPB). The AK-based measurements are TST, FTSS, and TUG which are also the components of the SPPB.
  Interventions: Diagnostic Test: Azure Kinect-based Tandem Stance Test (ATST) and Physical Therapist's Measurements of Tandem Stance Test (PTST); Diagnostic Test: Azure Kinect-based Five Times Sit-to-Stand Test (AFTSS) and Physical Therapist's Measurements of Five Times Sit-to-Stand Test (PFTSS); Diagnostic Test: Azure Kinect-based Timed Up and Go Test (ATUG) and Physical Therapist's Measurements of Timed Up and Go Test (PTUG); Diagnostic Test: Short Physical Performance Battery (SPPB); Diagnostic Test: Berg Balance Scale (BBS); Diagnostic Test: Functional Reach Test (FRT); Diagnostic Test: Four-Square Step Test (FSST); Diagnostic Test: Grip Strength (GS)

INTERVENTIONS:
Diagnostic Test: Azure Kinect-based Tandem Stance Test (ATST) and Physical Therapist's Measurements of Tandem Stance Test (PTST) — For the Tandem Stance Test comparisons, the Azure Kinect-based Tandem Stance Test system quantified the distance traveled by the pelvic point to X, Y, and Z coordinates over a 30-second duration while the physical therapist measured the time elapsed until the participant lost balance was measured with a maximum of 30 seconds. Participants remained a tandem stance, positioning their preferred leg in front such that the heel of the front foot touched the toes of the back foot, ensuring both feet were aligned as straight as possible. They stood with holding on to two chairs each placed on their sides for stability and safety. Upon the cue to 'start', the participants let their hands go and both the Azure Kinect-based system and the physical therapist's stopwatch initiated their measurements. Participants tried to maintain their stance for 30 seconds. The participants had to reposition themselves when they stepped, used hands or lose balance for 30 seconds
Diagnostic Test: Azure Kinect-based Five Times Sit-to-Stand Test (AFTSS) and Physical Therapist's Measurements of Five Times Sit-to-Stand Test (PFTSS) — The Five Times Sit-to-Stand Test (FTSS), standardized by Csuka and McCarty, has been designed to assessing lower limb strength as well as balance and postural control among elder population with high level of reliability. A previous study reported excellent intra-rater reliability (ICC=.914-.933) and inter-rater reliability (ICC=.988-.995) among healthy older adults. In addition, Five Times Sit-to-Stand Test more than 11.50 seconds had been reported to represent risk of falls among elders over 65-year-old. To assess Five Times Sit-to-Stand Test , a chair, 45cm in height and fixed to the ground, was placed three meters from the camera. Participants began seated, and on start cue, repeatedly stood up and sat down five times. The Azure Kinect-based system automatically ended its measurement as the participant completed the fifth stand, whereas the physical therapist manually measured time using the stopwatch. The time measures from the system and therapist were compared.
Diagnostic Test: Azure Kinect-based Timed Up and Go Test (ATUG) and Physical Therapist's Measurements of Timed Up and Go Test (PTUG) — The Timed Up and Go test (TUG) has been employed as a straightforward assessment of an individual's mobility, necessitating both static and dynamic balance. A Timed Up and Go test duration exceeding 9.50 seconds has been identified as indicative of a heightened fall risk in individuals aged 65 and older. A previous study reported excellent intra-rater reliability (ICC=.97) and inter-rater reliability (ICC=.96). Initiating in a seated position, participants stood upon commencement of the test. Simultaneously, the Azure Kinect-based system and stopwatch began the time measurements. Participants then walked a distance of three meters, turned around, retraced their steps, and resumed their seated position. The Azure Kinect-based system automatically terminated its timing once the participant was seated, while the physical therapist manually stopped the stopwatch. The time measures from the system and therapist were compared.
Diagnostic Test: Short Physical Performance Battery (SPPB) — The assessment includes three tests: a Timed Up and Go test test where participants walked a distance of 3 meters at their comfortable pace; a Five Times Sit-to-Stand Test which the duration is also measured; and the standing balance test which determines a participant's capacity to maintain three different stances of side-by-side, semi-tandem, and full tandem, each for 10 seconds.
Diagnostic Test: Berg Balance Scale (BBS) — Participants are scored on a 5-point scale for each task, where a score of 0 signifies an inability to perform, while a 4 denotes independence in execution. A perfect score of 56 is a marker of excellent balance. Administering the Berg Balance Scale is efficient, taking between 10 to 20 minutes, and requires only basic equipment such as a chair, stopwatch, ruler, and step within a small space.
Diagnostic Test: Functional Reach Test (FRT) — Participants, standing barefoot, aligned the side of their body with a wall, ensuring no contact. Their stance was parallel with feet comfortably spaced. With their shoulders flexed at a 90° angle adjacent to the wall, they kept their elbows straight and hands clenched. The starting point on a horizontally affixed measuring tape, level with the floor, was determined by where the third metacarpal touched. This tape was aligned with each participant's acromion height. Without taking a step, lifting heels or losing balance, participants leaned forward to their maximum extent. The difference between the initial and final third metacarpal positions on the tape denoted the reach distance.
Diagnostic Test: Four-Square Step Test (FSST) — During the Four-Square Step Test, participants were instructed to step over four straight tapes, each 90 cm in length, laid out in a cross-shape configuration on the floor. Beginning in square 1 and facing square 2, participants followed a specific sequence: they stepped forward into the next quadrant, then to the right, backward, and finally to the left, moving in a clockwise direction. This sequence was then retraced in a counterclockwise manner. It was essential for both feet to touch down in each quadrant. Participants aimed to complete this pattern as fast as they could, avoiding stepping the tapes. The duration taken to finish the sequence was recorded.
Diagnostic Test: Grip Strength (GS) — The strength of the dominant hand's maximal grip force, indicative of upper extremity muscle strength, was gauged using a digital isometric hand dynamometer.

SUMMARY:
Falls significantly reduce physical function as well as quality of life which leads to failure of successful aging among elders. There is a great need for automated assessing physical functions that can be address fall risks for those elderly living alone. The study aims to test validity and reliability of a depth camera-based physical function and fall risk assessment among healthy young and elderly adults with and without fall histories.

The present study explores the concurrent, convergent, and discriminative validity of Azure Kinect-based physical function assessments, along with the intra-rater and inter-rater reliability of these measurements. The diagnostic accuracy and the optimal cut-off values of the Azure Kinect-based tests in differentiating fall risks will be provided.

The enrolled participants will complete the following evaluations during a single session: Tandem Stance Test (TST), Five Times Sit to Stand Test (FTSS), Turn Up and Go Test (TUG), Berg Balance Scale (BBS), Functional Reach Test (FRT), Four Square Step Test (FSST), Grip Strength (GS), and Short Physical Performance Battery (SPPB). Each of the AK-based evaluation will be measured three times with simultaneous measurements of the same physical therapist directed tests: two trials will be measured by one physical therapist, while one trial will be measured by the another physical therapist.

ELIGIBILITY:
Inclusion Criteria:

* those who: (1) are adults (≥18 years); (2) are able to follow instructions during physical examinations; (3) can walk independently for at least six meters; and (4) agrees to participate and provide written consent.

Exclusion Criteria:

* those who have: (1) orthopedic injuries; (2) neurological disease; (3) pain or inflammation; (4) visual or hearing problems; (5) a previous history of surgery; (6) serious medical concerns; or (7) refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
AK-based Tandem Stance Test and Physical Therapist's Measurements of Tandem Stance Test | baseline
  For the Tandem Stance Test comparisons, the Azure Kinect-based Tandem Stance Test system quantifies the distance traveled by the pelvic point in X, Y, and Z coordinates over a 30-second duration, while the physical therapist measures the time elapsed until the participant loses balance, with a maximum of 30 seconds. Participants remain in a tandem stance, positioning their preferred leg in front so that the heel of the front foot touches the toes of the back foot, ensuring both feet are aligned as straight as possible. They stand holding onto two chairs placed on their sides for stability and safety. Upon the cue to 'start', the participants let go of their hands, and both the system and the physical therapist's stopwatch initiate measurements. Participants try to maintain their stance for 30 seconds. Repositioning is noted when they step, use hands, or lose balance before 30 seconds. The total displacement (meters) and time until losing balance (seconds) are measured.
AK-based Five Times Sit-to-Stand Test (AFTSS) and Physical Therapist's Measurements of Five Times Sit-to-Stand Test | baseline
  To assess Five Times Sit-to-Stand Test, a chair, 45cm in height and fixed to the ground, is placed three meters from the camera. Participants begin seated, and on start cue, repeatedly standd up and sit down five times. The Azure Kinect-based system automatically ends its measurement as the participant complete the fifth stand, whereas the physical therapist manually measures time using the stopwatch. The time measures in seconds from the system and therapist are compared.
AK-based Timed Up and Go Test and Physical Therapist's Measurements of Timed Up and Go Test | baseline
  The Timed Up and Go test measures a person's mobility requiring both static and dynamic balance. Testing initiates with the participant moving from sit to stand and progresses through walking three meters within the laboratory, turning around, retracing steps, and returning to sit. The Azure Kinect-based system automatically stops timing the instant the participant sits, as does the physical therapist, who uses a stopwatch. The time to complete the tasks are measured in seconds.

SECONDARY OUTCOMES:
Short Physical Performance Battery | baseline
  Short Physical Performance Battery is comprised of three tests: a Timed Up and Go test where the respondent walks a distance of 3 meters at their comfortable pace, a Five Times Sit to Stand test that also measures duration, and a standing balance test which determines a respondent's capacity to maintain three different stances of side-by-side, semi-tandem, and full tandem, each for 10 seconds.
  The time to complete each task are measured in seconds
Berg Balance Scale | baseline
  Participants are scored from 0-4 for each task, where a score of 0 indicates an inability to perform the task, while 4 denotes independence in execution. The maximal total score is 56, indicating that an individual has perfect balance. Administering the Berg Balance Scale is efficient, taking between 10 to 20 minutes, and requires only basic equipment such as a chair, a stopwatch, a ruler, and a step within a small space. The score in points are measured after completion of all tasks in the Berg Balance Scale.
Functional Reach Test | baseline
  Participants, standing without shoes on, place their side in a line with the wall so that there is no contact. Their stance is symmetrical with feet comfortably spaced. Their shoulders are flexed at a 90° angle to the wall, elbows remain extended, and fists are clenched. The zero point is established at the touch point of the third metacarpal on a horizontally mounted measuring tape, level with the floor. The tape is aligned with each participant's acromion height. Participants are then directed to reach forward maximally without taking a step, lifting their heels, or losing balance. The reach distance is measured as the difference between the initial and final third metacarpal positions on the tape. The distances of the reach are measured in meters.
Four-Square Step Test | baseline
  The subjects are instructed to step over four pieces of straight tape (90 cm long) arranged in a cross on the ground. The subjects step forward into the next quadrants, then to their right into the next quadrant, then backward to the last quadrant, and finally leftward into the starting quadrant, proceeding in a clockwise sequence. This pattern is then retraced in reverse order. Both feet must land in every quadrant. Subjects are instructed to perform this pattern as quickly as possible while trying not to step on the tapes. The time taken to complete this sequence is recorded in seconds
Grip Strength | baseline
  The maximal grip force strength of the dominant hand, representative of muscle strength in the upper extremity, is measured with a digital isometric hand dynamometer (Electronic hand dynamometer, PRO-SPECS®, Seoul, South Korea). The participant holds the shoulder adducted with the elbow flexed at 90° while keeping the forearm in a neutral position. The average from three attempts at squeezing is used for analysis. The grip strength are measured in weight (kilograms)

CONTACTS AND LOCATIONS:
Locations (1):
- Sahmyook University, Seoul, South Korea